CLINICAL TRIAL: NCT03191045
Title: Development of MRI Protocols to Assess Gastrointestinal Motility With Concomitant Perfused Manometry Validation in Healthy Volunteers
Brief Title: In Vivo Predictive Dissolution 1
Acronym: iPD1
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); University of Michigan (Other)
Responsible Party: Principal Investigator, Luca Marciani, Associate Professor, University of Nottingham
Other Study IDs: A14112016 MRI FDA
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: MRI; motility; perfused manometry; stomach; bowel; water
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: A group of 21 healthy adult participants studied twice (test-retest)
  Interventions: Diagnostic Test: MRI and concomitant perfused manometry of bowel motility

INTERVENTIONS:
Diagnostic Test: MRI and concomitant perfused manometry of bowel motility — We will carry out serial cine MRI of the bowel. At the same time we will record perfused manometry readings of the bowel in healthy adult participants.

SUMMARY:
This study will: 1. validate MRI motility method with concomitant perfused manometry method in healthy adult participants. 2. measure exploratory endpoints of interest including GI fluid volumes in 21 adult healthy volunteers studied twice.

DETAILED DESCRIPTION:
The gastrointestinal (GI) environment where drug products dissolve has not been studied in detail due to limitations, especially invasiveness of existing techniques. Hence little in vivo data on GI fluids and motility is available to improve relevance of predictive dissolution models and bench dissolution techniques. Recent advances in magnetic resonance imaging (MRI) methods could provide novel data and insights. On-going studies at the University of Michigan and at the University of Nottingham, using advanced, validated, quantitative MRI techniques have already shown that GI fluid (water) volumes can be measured. The classical method for measuring GI motility is via a manometric method involving intubation, but it is possible to measure GI motility with MRI. Based on our MRI motility pilot data and on the literature available, this study aims to test the main hypotheses that in healthy adult participants the new MRI method has the potential to replace current manometric study protocols and will allow a simultaneous measurement of gastrointestinal motility and fluid volumes in the gut during the fasted state. This will establish a solid and unprecedented base of in vivo results upon which to base advances in oral pharmaceutical product science. For this initial study, the study objectives are therefore: 1. To validate the MRI motility method with concomitant perfused manometry method in healthy adult participants. 2. To measure exploratory endpoints of interest including GI fluid volumes. Twenty one adult healthy volunteers will participate in this replicated study. We will pass a thin perfused manometry tube via the nose into the gut of the participants and then take MRI images of abdominal areas while bowel motility is being measured via a tube manometric method to see how they compare. We will be able also to measure the volume of fluids in the gut.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60
* Healthy
* Male or female
* Able to give informed written consent and willing to comply with required study procedures

Exclusion Criteria:

* Any history of serious, unstable medical condition, unstable/uncontrolled diabetes mellitus, and/ or major psychiatric diagnosis such as attention deficit hyperactivity disorder, obsessive compulsive disorder, panic attacks and generalized anxiety disorder.
* Any reported history of gastrointestinal disease
* Any significant respiratory disease such as asthma
* Any conditions requiring daily intake of any prescription and/or over-the-counter medications
* Any reported history of surgery that could affect gastrointestinal function (e.g. colectomy, small bowel resection)
* Reported alcohol dependence
* Abnormal screening procedures and laboratory results that are clinically significant in the opinion of the study medically qualified researcher
* Pregnancy
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Inability to lie flat
* Weight exceeding scanner limits of 120kg
* Poor understanding of English language
* Any conditions causing fidgeting
* Claustrophobia
* Participation of any medical trials for the past 3 months
* Judgement by the study medically qualified researcher that the candidate will be unable to comply with the full study protocol e.g. severe chronic obstructive pulmonary disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Self-reporting, healthy adult participants, with no restrictions on gender, ethnicity or race, recruited by advertisement by poster and flyer
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Stomach MRI motility | Over set time bins and recorded for up to 4 hours
  Area under the curve (AUC) of the stomach motility contractions (in mm×second) measured by MRI.

SECONDARY OUTCOMES:
Stomach perfused manometry motility | Over set time bins and recorded for up to 4 hours
  Area under the curve (AUC) of the stomach motility contractions (in mmHg×second) measured by perfused manometry

OTHER OUTCOMES:
Stomach MRI and perfused manometry correlation | Over set time bins and recorded for up to 4 hours
  Correlation between the area under the curves (AUCs) of the MRI and perfused manometry stomach motility contractions
Small bowel MRI motility | Over set time bins and recorded for up to 4 hours
  Small bowel motility by MRI (both in arbitrary units and, where possible, using actual diameter readings as above in mm×second)
Small bowel perfused manometry motility | Over set time bins and recorded for up to 4 hours
  Small bowel motility by perfused manometry (as above, in mmHg×second)
Small bowel MRI and perfused manometry correlation | Over set time bins and recorded for up to 4 hours
  Correlation between the area under the curves (AUCs) of the MRI and perfused manometry small bowel motility contractions
Bowel liquid volumes | Recorded for up to 4 hours
  Gastric, small bowel water and colonic freely mobile liquid volumes (in mL)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marciani, PhD, Principal Investigator — University of Nottingham; Gordon L Amidon, PhD, Principal Investigator — University of Michigan; Greg E Amidon, PhD, Principal Investigator — University of Michigan; Maura Corsetti, MD, Principal Investigator — University of Nottingham; Jeff Wright, PhD, Principal Investigator — University of Nottingham; Paul Glover, PhD, Principal Investigator — University of Nottingham; Geoffrey S Hebbard, PhD, Principal Investigator — Melbourne Health; Caroline L Hoad, PhD, Principal Investigator — University of Nottingham; Penny A Gowland, PhD, Principal Investigator — University of Nottingham; Kerby Shedden, PhD, Principal Investigator — University of Michigan; Joseph Dickens, PhD, Principal Investigator — University of Michigan; Robin C Spiller, MD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Digestive Diseases Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heissam K, Abrehart N, Hoad CL, Wright J, Menys A, Murray K, Glover PM, Hebbard G, Gowland PA, Baker J, Hasler WL, Spiller RC, Corsetti M, Brasseur JG, Hens B, Shedden K, Dickens J, Mudie DM, Amidon GE, Amidon GL, Marciani L. Measurement of fasted state gastric antral motility before and after a standard bioavailability and bioequivalence 240 mL drink of water: Validation of MRI method against concomitant perfused manometry in healthy participants. PLoS One. 2020 Nov 11;15(11):e0241441. doi: 10.1371/journal.pone.0241441. eCollection 2020. PMID 33175860